CLINICAL TRIAL: NCT03326921
Title: Phase I Study of Adoptive Immunotherapy With CD8+ and CD4+ Memory T Cells Transduced to Express an HA-1-Specific T Cell Receptor (TCR) for Children and Adults With Recurrent Acute Leukemia After Allogeneic Hematopoietic Stem Cell Transplantation (HCT)
Brief Title: HA-1 T TCR T Cell Immunotherapy for the Treatment of Patients With Relapsed or Refractory Acute Leukemia After Donor Stem Cell Transplant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: HighPass Bio, Inc. (Unknown); PromiCell Therapeutics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9716; NCI-2017-01054 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9716 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9217022 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-10-05; First posted 2017-10-31 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Juvenile Myelomonocytic Leukemia; Recurrent Acute Biphenotypic Leukemia; Recurrent Acute Undifferentiated Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Refractory Acute Lymphoblastic Leukemia; Refractory Adult Acute Lymphoblastic Leukemia; Blast Phase Chronic Myeloid Leukemia, BCR-ABL1 Positive; Recurrent Blastic Plasmacytoid Dendritic Cell Neoplasm; Recurrent Myelodysplastic Syndrome; Refractory Blastic Plasmacytoid Dendritic Cell Neoplasm; Refractory Myelodysplastic Syndrome; Acute Undifferentiated Leukemia; Mixed Phenotype Acute Leukemia; Recurrent Chronic Myeloid Leukemia, BCR-ABL1 Positive; Refractory Chronic Myeloid Leukemia, BCR-ABL1 Positive; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Myelodysplastic Syndrome; Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Acute Biphenotypic Leukemia; Chronic Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Minimal Residual Disease; Recurrent Chronic Myelomonocytic Leukemia; Recurrent Mixed Phenotype Acute Leukemia; Leukemia; Chronic Myeloid Leukemia, BCR-ABL1 Positive
Keywords: HA-1; TCR; Immunotherapy; Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Juvenile; Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Blastic Plasmacytoid Dendritic Cell Neoplasm; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Neoplasm, Residual; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CD4+ and CD8+ HA-1 TCR T cells) (Experimental): Patients receive lymphodepleting chemotherapy (e.g., fludarabine and cyclophosphamide or debulking regimens as specified in the protocol) ending 2-14 days prior to HA-1 TCR T cell administration. Patients then receive CD4+ and CD8+ HA-1 TCR T cells IV.
  Interventions: Biological: CD8+ and CD4+ Donor Memory T-cells-expressing HA1-Specific TCR; Procedure: Bone Marrow Aspiration; Procedure: Biospecimen Collection

INTERVENTIONS:
Biological: CD8+ and CD4+ Donor Memory T-cells-expressing HA1-Specific TCR — Given IV
  Other Names: CD8+ and CD4+ Donor Memory T-cells-expressing pRRLSIN iC9-HA1 TCR2-RQR-CD8; HA-1 TCR CD8+ and CD4+ Tm Cells; HA-1 TCR T Cells
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection

SUMMARY:
This phase I trial studies the side effects and best dose of CD4+ and CD8+ HA-1 T cell receptor (TCR) (HA-1 T TCR) T cells in treating patients with acute leukemia that persists, has come back (recurrent) or does not respond to treatment (refractory) following donor stem cell transplant. T cell receptor is a special protein on T cells that helps them recognize proteins on other cells including leukemia. HA-1 is a protein that is present on the surface of some peoples' blood cells, including leukemia. HA-1 T cell immunotherapy enables genes to be added to the donor cells to make them recognize HA-1 markers on leukemia cells.

DETAILED DESCRIPTION:
OUTLINE:

This is a dose-escalation study of CD4+ and CD8+ HA-1 TCR T cells.

Patients receive lymphodepleting chemotherapy (e.g., fludarabine and cyclophosphamide or debulking regimens as specified in the protocol) ending 2-14 days prior to HA-1 TCR T cell administration. Patients then receive CD4+ and CD8+ HA-1 TCR T cells intravenously (IV).

After completion of study treatment, patients are followed up closely for 12 weeks and then every 6 months for years 1-5, and every year for years 6-15.

Initial study activity was funded in part by HighPass Bio, Inc. Current study activity is funded in part by PromiCell Therapeutics, Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject age 0-80 years at the time of enrollment.
* Subject must express HLA-A*0201
* Subject must have the HA-1(H) genotype (RS_1801284: A/G, A/A)
* Subject must have an adult donor for HCT who is adequately HLA matched by institutional standards (includes HLA-matched related or unrelated donors, and HLA-mismatched family donors, including haploidentical donors) and is either:

  * HLA-A*0201 positive and HA-1(H) negative (RS_1801284: G/G) or
  * HLA-A*0201 negative
* Subjects who are currently undergoing or who previously underwent allogeneic HCT for

  * Acute myeloid leukemia (AML) of any subtype
  * Acute lymphoid leukemia (ALL) of any subtype
  * Mixed phenotype/undifferentiated/any other type of acute leukemia, including blastic plasmacytoid dendritic cell neoplasm
  * Chronic myeloid leukemia with a history of blast crisis and:

    * With relapse or refractory disease (>= 5% marrow blasts, or circulating blasts) at any time after HCT
    * With persistent rising minimal residual disease (defined as detectable disease by morphology, flow cytometry, molecular or cytogenetic testing but < 5% marrow blasts by morphology, no circulating blasts on >= 2 of two consecutive tests), refractory or ineligible for treatment with tyrosine kinase inhibitors at any time after HCT
  * Myelodysplastic syndrome (MDS) of any subtype
  * Chronic myelomonocytic leukemia (CMML)
  * Juvenile myelomonocytic leukemia (JMML)
* Subjects must be able to understand and be willing to give informed consent; decision-impaired adults may consent with their legally authorized representative; parent or legal representative will be asked to consent for subjects younger than 18 years old
* Subjects must agree to participate in long-term follow-up for up to 15 years if they are enrolled in the study and receive T cell infusion
* Subjects who have relapsed or have MRD after HCT may receive other agents for treatment of disease and remain eligible for the protocol
* A specific performance status score is not required for enrolling on the protocol; a delay in infusion of the HA-1 TCR T cells may be required for subjects with low performance status

DONOR SELECTION INCLUSION

* Donor age >= 18 years
* Donors must be able to give informed consent

Exclusion Criteria:

* Medical or psychological conditions that would make the subject unsuitable candidate for cell therapy at the discretion of the principal investigator (PI)
* Fertile subjects unwilling to use contraception during and for 12 months after treatment
* Subjects with a life expectancy of < 3 months of enrollment from coexisting disease other than leukemia
* Subjects who have ongoing grade IV acute GVHD or severe chronic GVHD following most recent transplant. Exception: the principal investigator (PI) may make an exception on a case-by-case basis to include such a subject if there is doubt surrounding the GVHD diagnosis and/or sustained significant improvement in GVHD severity
* The presence of organ toxicities will not necessarily exclude subjects from enrolling on the protocol at the discretion of the PI; however, a delay in the infusion of HA-1 TCR T cells may be required

DONOR SELECTION EXCLUSION

* Donors who are human immunodeficiency virus (HIV)-1, HIV-2, human T-lymphotropic virus (HTLV)-1, HTLV-2 seropositive or with active hepatitis B or hepatitis C virus infection
* Unrelated donor residing outside of the United States of America (USA) unless the donor screening, testing and leukapheresis occur at an National Marrow Donor Program (NMDP)-affiliated and qualified donor center and are facilitated by the NMDP

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2027-10-16 (Estimated); Study Completion 2028-07-16 (Estimated)

PRIMARY OUTCOMES:
Feasibility of manufacturing minor H antigen (HA-1) T cell receptor (TCR) CD8+ and CD4+ T cells | At time of T cell infusion (at day 0)
  Proportion of subjects for whom a HA-1 TCR T cell product can be produced.
Feasibility of administering minor H antigen (HA-1) T cell receptor (TCR) CD8+ and CD4+ T cells | At time of T cell infusion (at day 0)
  Proportion of subjects for whom a HA-1 TCR T cell product can be administered.
Incidence of dose-limiting toxicities of HA-1 T cell receptor (TCR) T cells | Up to 12 weeks after T-cell infusion
  Toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.

SECONDARY OUTCOMES:
Duration of in vivo persistence of transferred HA-1 T cell receptor (TCR) CD4+ T cells in peripheral blood | Up to 1 year
  Evaluated by tetramer and/or molecular tracking e.g. quantitative polymerase chain reaction (qPCR).
Duration of in vivo persistence of transferred HA-1 T cell receptor (TCR) CD8+ T cells in peripheral blood | Up to 1 year
  Evaluated by tetramer and/or molecular tracking e.g. qPCR.
Presence, proportion and persistence of HA-1 T cell receptor (TCR) CD4+ T cells in the bone marrow | Up to 1 year
  Evaluated by tetramer and/or molecular tracking e.g. qPCR.
Presence, proportion and persistence of HA-1 T cell receptor (TCR) CD8+ T cells in the bone marrow | Up to 1 year
  Evaluated by tetramer and/or molecular tracking e.g. qPCR.
Specific cytolytic activity of HA-1 T cell receptor (TCR) CD8+ and CD4+ T cells against HLA-A*0201+ HA-1+ target cells before adoptive T cell transfer | At the time of T cell infusion (at day 0)
  Assessed by in vitro chromium release assay or equivalent cytotoxicity assay.
Specific cytolytic activity of HA-1 T cell receptor (TCR) CD8+ and CD4+ T cells against HLA-A*0201+ HA-1+ target cells after adoptive T cell transfer | Up to 1 year
  By in vitro chromium release assay or flow cytometric degranulation assay (CD107a) using samples of peripheral blood and/or bone marrow collected from subjects after adoptive T cell transfer.
Reduction of leukemia in the bone marrow in subjects who have measurable leukemia in the marrow prior to HA-1 T cell receptor (TCR) T cell infusion | Up to 1 year
  Quantified by flow cytometry to determine percentage of leukemic cells in the marrow.
Reduction of recipient normal hematopoietic cells in the bone marrow in subjects who have measurable recipient normal hematopoietic cells in the marrow prior to HA-1 T cell receptor (TCR) T cell infusion | Up to 1 year
  Quantified by variable number tandem repeat (VNTR) to determine percentage of normal recipient and donor cells in the marrow.
Proportion of subjects who develop new or recurrent symptoms or signs of graft-versus-host disease | Up to 1 year
  Assessed using clinical evaluation and standard clinical graft versus host disease (GVHD) grading criteria

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Krakow, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krakow EF, Brault M, Summers C, Cunningham TM, Biernacki MA, Black RG, Woodward KB, Vartanian N, Kanaan SB, Yeh AC, Dossa RG, Bar M, Cassaday RD, Dahlberg A, Till BG, Denker AE, Yeung CCS, Gooley TA, Maloney DG, Riddell SR, Greenberg PD, Chapuis AG, Newell EW, Furlan SN, Bleakley M. HA-1-targeted T-cell receptor T-cell therapy for recurrent leukemia after hematopoietic stem cell transplantation. Blood. 2024 Sep 5;144(10):1069-1082. doi: 10.1182/blood.2024024105. PMID 38683966